CLINICAL TRIAL: NCT03445728
Title: Effects of Nicorandil on Cardiac Infarct Size in Patients With ST-segment Elevation Acute Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: China-Administration of Nicorandil Group（CHANGE）
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: First People's Hospital of Yulin (Other); Beijing Chao Yang Hospital (Other); Wuhan Asia Heart Hospital (Other); Hainan Hospital of PLA General Hospital (Unknown); Zunyi Medical College (Other); Guizhou Provincial People's Hospital (Other); Second Affiliated Hospital of Nanchang University (Other); The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yun Dai Chen, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHANGE 001
Record Dates: First submitted 2018-02-02; First posted 2018-02-26 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Infarction; Percutaneous Coronary Intervention; Nicorandil
Keywords: Cardiac magnetic resonance; Infarct Size
MeSH Terms: conditions — Myocardial Infarction | interventions — Nicorandil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Patients were randomly assigned to two groups before emergent coronary angiography: those who received intravenous (iv.) nicorandil before and after (ivgtt.) reperfusion with PCI (nicorandil group);
  Interventions: Drug: Nicorandil
- Placebo arm (Placebo Comparator): Patients were randomly assigned to two groups before emergent coronary angiography, those who received placebo before and after reperfusion with PCI.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicorandil — After randomization, receive primary PCI and standard therapy, 12mg Nicorandil iv. just before ballooning or stenting, then keep Nicorandil 6mg/h ivgtt. up to 24h
  Arms: Treatment arm
Other: Placebo — After randomization, receive primary PCI and standard therapy, just like the intervension group also iv. just before ballooning or stenting, then keep ivgtt. up to 24h
  Arms: Placebo arm

SUMMARY:
We compared the infarct size in ST-segment elevation myocardial infarction (STEMI) patients undergoing primary percutaneous coronary intervention (PCI) treated by nicorandil before and after the reperfusion with those standard therapy treated by PCI

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of nicorandil in improving myocardial infarct size in patients with acute myocardial infarction through a multi-center, prospective, randomized, double-blind and parallel-controlled clinical study, providing evidence-based support for the optimization of PCI treatment strategies. The primary objective of the study was to compare whether the effect of nicorandil in combination with PCI was significantly better at reducing the myocardial infarct size than that of PCI alone in AMI patients.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ST-T elevation MI patients (<12h)
2. undergoing emergency PCI；
3. Subject has read and signed a written, informed consent form.

Exclusion Criteria:

1. SBP<80mmHg；
2. LM stenosis
3. Aortic dissection；
4. AMI (<6 month)
5. PCI或CABG (<6 month)
6. Already under the treatment of Nicorandil；
7. Contraindicated or intolerable to Nicorandil
8. severe adverse effects to CMR or MRI；
9. Currently (or within one month) participating in another new drug trial.；
10. Pregnant or lactation period；
11. Severe somatic disease preventing the participant from completing the trial, or based on the discretion of the investigators, the patient is incapable of participating; Individuals with abnormal laboratory test results and/or clinical manifestations rendering them unsuitable to participate as judged by the investigators;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Infarct size as measured by cardiac MRI | 7 days after primary PCI
  The myocardial infarct size was derived by measuring the area of delay-enhanced image-enhanced MRI, which was judged and analyzed by two experienced MRI cardiac diagnosticians.

SECONDARY OUTCOMES:
Infarct size as measured by cardiac MRI | 6 months after PCI
  The myocardial infarct size was derived from the program's automatic analysis of delayed enhancement images.
Corrected thrombolysis in myocardial infarction (TIMI) frame count (cTFC) | 5 minutes after stent implantation during PCI
  the starting point is the number of frames in which the contrast agent completely or nearly completely filled the beginning of the coronary artery and touched both sides of the coronary vessel wall, and the end point is the number of frames in which the contrast agent entered the distal branch vessel and developed a specific anatomical marker
Incidence of slow flow/no-reflow | 5 minutes after stent implantation during PCI
  When scanning at a rate of 15 frames per second, cTFC > 27 frames per second was used as the criterion for the diagnosis of slow blood flow after primary PCI
ST-segment fall rate of electrocardiogram (ECG) | 2 hours after the procedure
  Complete ST-segment resolution at 2 h after PCI
Serum creatinine kinase (CK-MB) level | Baseline, 6, 12, 18, 24 hours after the PCI
  Change of serum creatinine kinase
Edema size (LV area %) measured by cardiac MRI | 7 days after the procedure
  Edema size
Microvascular obstructionmeasured by cardiac MRI | 7 days after the procedure
  Microvascular obstructionmeasured
LV Ejection fraction (%) as measured by cardiac MRI | 7 days after the procedure
  LV Ejection fraction in early phase
LV Ejection fraction (%) as measured by cardiac MRI | 6 months after the procedure
  LV Ejection fraction in late phase
MACE | up to 12 months
  all-cause death, cardiovascular death, , Rehospitalization for heart failure, Unplanned PCI After PPCI
CIN | 48-72 hours after primary PCI
  contrast induced nephropathy

CONTACTS AND LOCATIONS:
Overall Officials: Yundai Chen, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- CHINA, Beijing, China

REFERENCES:
- [Result] Ishii H, Ichimiya S, Kanashiro M, Amano T, Imai K, Murohara T, Matsubara T. Impact of a single intravenous administration of nicorandil before reperfusion in patients with ST-segment-elevation myocardial infarction. Circulation. 2005 Aug 30;112(9):1284-8. doi: 10.1161/CIRCULATIONAHA.104.530329. Epub 2005 Aug 22. PMID 16116055
- [Result] Ito H, Taniyama Y, Iwakura K, Nishikawa N, Masuyama T, Kuzuya T, Hori M, Higashino Y, Fujii K, Minamino T. Intravenous nicorandil can preserve microvascular integrity and myocardial viability in patients with reperfused anterior wall myocardial infarction. J Am Coll Cardiol. 1999 Mar;33(3):654-60. doi: 10.1016/s0735-1097(98)00604-4. PMID 10080465
- [Result] Kitakaze M, Asakura M, Kim J, Shintani Y, Asanuma H, Hamasaki T, Seguchi O, Myoishi M, Minamino T, Ohara T, Nagai Y, Nanto S, Watanabe K, Fukuzawa S, Hirayama A, Nakamura N, Kimura K, Fujii K, Ishihara M, Saito Y, Tomoike H, Kitamura S; J-WIND investigators. Human atrial natriuretic peptide and nicorandil as adjuncts to reperfusion treatment for acute myocardial infarction (J-WIND): two randomised trials. Lancet. 2007 Oct 27;370(9597):1483-93. doi: 10.1016/S0140-6736(07)61634-1. PMID 17964349
- [Result] Bulluck H, Hammond-Haley M, Weinmann S, Martinez-Macias R, Hausenloy DJ. Myocardial Infarct Size by CMR in Clinical Cardioprotection Studies: Insights From Randomized Controlled Trials. JACC Cardiovasc Imaging. 2017 Mar;10(3):230-240. doi: 10.1016/j.jcmg.2017.01.008. PMID 28279370
- [Result] Ishii H, Ichimiya S, Kanashiro M, Amano T, Ogawa Y, Mitsuhashi H, Sakai S, Uetani T, Murakami R, Naruse K, Murohara T, Matsubara T. Effect of intravenous nicorandil and preexisting angina pectoris on short- and long-term outcomes in patients with a first ST-segment elevation acute myocardial infarction. Am J Cardiol. 2007 May 1;99(9):1203-7. doi: 10.1016/j.amjcard.2006.12.034. Epub 2007 Mar 16. PMID 17478142
- [Result] IONA Study Group. Effect of nicorandil on coronary events in patients with stable angina: the Impact Of Nicorandil in Angina (IONA) randomised trial. Lancet. 2002 Apr 13;359(9314):1269-75. doi: 10.1016/S0140-6736(02)08265-X. PMID 11965271
- [Result] Okamura A, Rakugi H, Ohishi M, Yanagitani Y, Shimizu M, Nishii T, Taniyama Y, Asai T, Takiuchi S, Moriguchi K, Ohkuro M, Komai N, Yamada K, Inamoto N, Otsuka A, Higaki J, Ogihara T. Additive effects of nicorandil on coronary blood flow during continuous administration of nitroglycerin. J Am Coll Cardiol. 2001 Mar 1;37(3):719-25. doi: 10.1016/s0735-1097(00)01171-2. PMID 11693742
- [Result] Kostic J, Djordjevic-Dikic A, Dobric M, Milasinovic D, Nedeljkovic M, Stojkovic S, Stepanovic J, Tesic M, Trifunovic Z, Zamaklar-Tifunovic D, Radosavljevic-Radovanovic M, Ostojic M, Beleslin B. The effects of nicorandil on microvascular function in patients with ST segment elevation myocardial infarction undergoing primary PCI. Cardiovasc Ultrasound. 2015 May 27;13:26. doi: 10.1186/s12947-015-0020-9. PMID 26012474
- [Derived] Qian G, Zhang Y, Dong W, Jiang ZC, Li T, Cheng LQ, Zou YT, Jiang XS, Zhou H, A X, Li P, Chen ML, Su X, Tian JW, Shi B, Li ZZ, Wu YQ, Li YJ, Chen YD. Effects of Nicorandil Administration on Infarct Size in Patients With ST-Segment-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: The CHANGE Trial. J Am Heart Assoc. 2022 Sep 20;11(18):e026232. doi: 10.1161/JAHA.122.026232. Epub 2022 Sep 8. PMID 36073634